CLINICAL TRIAL: NCT01881672
Title: Syndrome and Aspiration Pneumonia in Intensive Care
Acronym: SPIRE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Other Study IDs: SPIRE
Record Dates: First submitted 2013-06-13; First posted 2013-06-20 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: ICU Patients; Under Mechanical Ventilation; In State of Coma (Define by Glasgow ≤ 8); No Antibiotic Treatment
Keywords: Aspiration pneumonia; Coma; Mechanical ventilation
MeSH Terms: conditions — Pneumonia, Aspiration; Coma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Coma patients in ICU under mechanical ventilation

SUMMARY:
Inhalation is a common condition in patients with impaired their awareness requiring protection of the upper airway by endotracheal intubation. This inhalation may lead to chemical pneumonitis and/or bacterial pneumonia. Only the latter requires the administration of antibiotics. Patients developing such a bacterial pneumonia, has a mortality, duration of mechanical ventilation and length of ICU stay increased. However, the proportion of patients with such bacterial pneumonia, bacterial ecology and morbidity that are little known.

The aim of this study is to determine the frequency of bacterial pneumonia in patients admitted to the ICU for coma and treated with mechanical ventilation

ELIGIBILITY:
Inclusion Criteria:

* Altered consciousness defined by a Glasgow Coma Scale score less than or equal to 8 before protection of the upper airway by endotracheal intubation
* Patient under mechanical ventilation

Exclusion Criteria:

* Patient with pre-existing impairment of laryngeal function in Parkinson's disease, Alzheimer's disease, amyotrophic lateral sclerosis, laryngeal cancer, radiotherapy laryngeal
* Patient under guardianship
* Inpatient without consent
* Pregnant woman
* Patient previously treated with antibiotics for more than 24 hours at the time of ICU admission
* Patient with infection at ICU admission which justified probabilist antibiotic treatment
* Lack of social security
* Refusal of the patient or their next of kind

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in ICU for coma (define by Glasgow score < 8) and under mechanical ventilation. Suspicion of bacterial inhalation pneumonia will be confirme by a protected distal sampling during a flexible bronchoscopy.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2012-11; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Determine the frequency of bacterial pneumonia in patients admitted to the ICU for coma and treated with mechanical ventilation | ICU Discharge
  Participants will be followed for the duration of ICU stay, an expected average of 4 days

SECONDARY OUTCOMES:
Quantify the use of antibiotics during the ICU stay for patients admitted to the ICU for coma and treated with mechanical ventilation | ICU Discharge
  Participants will be followed for the duration of ICU stay, an expected average of 4 days
Description of the bacterial flora identified in respiratory specimens. | ICU Discharge
  Participants will be followed for the duration of ICU stay, an expected average of 4 days
Identification of predictive factors for development of bacterial pneumonia | ICU Discharge
  Participants will be followed for the duration of ICU stay, an expected average of 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Jean Baptiste Lascarrou, MD, Principal Investigator — CHD Vendee
Locations (1):
- CHD Vendee, La Roche-sur-Yon, France